CLINICAL TRIAL: NCT06780137
Title: A Phase 1b/2 Open-Label Clinical Study to Evaluate the Safety and Efficacy of MK-6070 and Ifinatamab Deruxtecan (I-DXd) in Participants With Relapsed/Refractory Extensive-Stage Small Cell Lung Cancer
Brief Title: A Study to Evaluate the Safety and Efficacy of Gocatamig (MK-6070) and Ifinatamab Deruxtecan (I-DXd) in Participants With Relapsed/Refractory Extensive-Stage Small Cell Lung Cancer (MK-6070-002)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6070-002; 2024-517926-25-00 (Registry Identifier: EU CT); MK-6070-002 (Other: MSD); jRCT2031250039 (Registry Identifier: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — durvalumab

STUDY DESIGN:
Intervention Model Description: Part 1 consists of four arms (gocatamig and I-DXd at different dosing intervals). Participants will be randomized to one of the four arms using an interactive response technology (IRT) system. Part 2 consist of three arms (gocatamig monotherapy in participants in Japan, gocatamig monotherapy in participants in China, and gocatamig at different dosing intervals). Part 3 consists of a single arm (gocatamig and durvalumab).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part 1 Arm 1: Gocatamig and I-DXd (Experimental): Participants will receive gocatamig and I-DXd at a determined dose until documented disease progression or discontinuation criteria are met.
  Interventions: Biological: Gocatamig; Biological: Ifinatamab Deruxtecan (I-DXd)
- Part 1 Arm 2: Gocatamig and I-DXd (Experimental): Participants will receive gocatamig and I-DXd at a determined dose until documented disease progression or discontinuation criteria are met.
  Interventions: Biological: Gocatamig; Biological: Ifinatamab Deruxtecan (I-DXd)
- Part 1 Arm 3a: I-DXd Monotherapy (Experimental): Participants will receive I-DXd until documented disease progression or discontinuation criteria are met.
  Interventions: Biological: Ifinatamab Deruxtecan (I-DXd)
- Part 1 Arm 3b: Gocatamig and I-DXd (Experimental): Participants will receive gocatamig and I-DXd at a determined dose until documented disease progression or discontinuation criteria are met.
  Interventions: Biological: Gocatamig; Biological: Ifinatamab Deruxtecan (I-DXd)
- Part 2 Arm 4: Gocatamig Monotherapy in Japan (Experimental): Participants in Japan will receive escalating doses of gocatamig until documented disease progression or discontinuation criteria are met.
  Interventions: Biological: Gocatamig
- Part 2 Arm 5: Gocatamig Monotherapy in China (Experimental): Participants in China will receive escalating doses of gocatamig until documented disease progression or discontinuation criteria are met.
  Interventions: Biological: Gocatamig
- Part 2 Arm 6: Gocatamig (Experimental): Participants will receive gocatamig at a determined dose until documented disease progression or discontinuation criteria are met.
  Interventions: Biological: Gocatamig
- Part 3 Arm 7: Gocatamig and Durvalumab (Experimental): Participants will receive gocatamig and durvalumab at a determined dose until documented disease progression or discontinuation criteria are met.
  Interventions: Biological: Gocatamig; Biological: Durvalumab

INTERVENTIONS:
Biological: Gocatamig — IV infusion
  Other Names: HPN328; MK-6070
  Arms: Part 1 Arm 1: Gocatamig and I-DXd; Part 1 Arm 2: Gocatamig and I-DXd; Part 1 Arm 3b: Gocatamig and I-DXd; Part 2 Arm 4: Gocatamig Monotherapy in Japan; Part 2 Arm 5: Gocatamig Monotherapy in China; Part 2 Arm 6: Gocatamig; Part 3 Arm 7: Gocatamig and Durvalumab
Biological: Ifinatamab Deruxtecan (I-DXd) — IV infusion
  Other Names: DS-7300a; MK-2400
  Arms: Part 1 Arm 1: Gocatamig and I-DXd; Part 1 Arm 2: Gocatamig and I-DXd; Part 1 Arm 3a: I-DXd Monotherapy; Part 1 Arm 3b: Gocatamig and I-DXd
Biological: Durvalumab — IV infusion
  Arms: Part 3 Arm 7: Gocatamig and Durvalumab

SUMMARY:
Researchers are looking for new ways to treat people with extensive-stage small cell lung cancer (SCLC) that has relapsed or is refractory. Gocatamig is a new type of immunotherapy that uses a person's immune system to find and destroy cancer cells. Ifinatamab deruxtecan (also known as I-DXd) is a drug which binds to a specific target on cancer cells and delivers treatment to destroy those cells. Durvalumab is a different type of immunotherapy that also destroys cancer cells. Researchers want to know if giving gocatamig, I-DXd, and gocatamig with I-DXd or durvalumab can treat SCLC that did not respond or stopped responding to a prior treatment.

The goals of this study are to learn:

* If gocatamig alone, I-DXd alone, and gocatamig with I-DXd or durvalumab are safe and well tolerated
* If people who receive gocatamig alone, I-DXd alone, and gocatamig with I-DXd or durvalumab have their SCLC get smaller or go away

DETAILED DESCRIPTION:
This study will consist of two parts. Part 1 will assess the safety, tolerability, and efficacy of gocatamig and I-DXd at doses determined in study MK-6070-001 (NCT: NCT04471727). Part 2 will assess the safety and tolerability of gocatamig in participants in Japan and China. Part 3 will assess the safety, tolerability, and efficacy of gocatamig with durvalumab.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically or cytologically confirmed SCLC that is extensive stage (defined as Stage IV (T any, N any, M1a/b/c) following at least 1 prior line of systemic therapy that included platinum-based chemotherapy
* Must be able to provide archival tumor tissue sample or fresh biopsy tissue sample
* Human immunodeficiency virus (HIV) infected participants must have well controlled HIV on antiretroviral therapy (ART)

Exclusion Criteria:

* Pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedure
* History of (noninfectious) pneumonitis/interstitial lung disease (ILD) that required steroids or has current pneumonitis/ILD, and or suspected ILD/pneumonitis
* Has clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses
* Active or history of immune deficiency with the exception of HIV-infected participants with well controlled HIV on ART
* History within 6 months before the first dose of study intervention of coronary/peripheral artery bypass graft and/or any coronary/peripheral angioplasty or clinically significant cardiovascular disease such as myocardial infarction, symptomatic congestive heart failure (CHF) (New York Heart Association > class II), and/or uncontrolled cardiac arrhythmia
* History of arterial thrombosis (eg, stroke or transient ischemic attack) within 6 months before the first dose of study intervention
* Active clinically significant infection requiring systemic therapy
* History of allogeneic tissue/solid organ transplant
* History of leptomeningeal disease
* Received prior radiotherapy within 2 weeks of start of study intervention, or has radiation-related toxicities, requiring corticosteroids
* Receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of chronic immunosuppressive therapy within 7 days prior to the first dose of study intervention
* Known additional malignancy that is progressing or has required active treatment within the past 3 years
* Untreated or symptomatic brain metastases
* Active viral hepatitis, defined as hepatitis A (hepatitis A virus immunoglobulin M [IgM] positive in the setting of associated signs/symptoms), hepatitis B (hepatitis B virus surface antigen [HbsAg] positive and/or detectable hepatitis B virus [HBV] deoxyribonucleic acid [DNA]), or hepatitis C (hepatitis C virus [HCV] antibody positive and detectable HCV ribonucleic acid). Participants with HBV with undetectable viral load after treatment are eligible. Participants with HCV with undetectable virus after treatment are eligible.
* Part 1 only: Radiation therapy to the lung >30 Gy within 6 months before the start of study intervention
* Part 1 only: Abdominal radiation within 4 weeks before start of study intervention
* Part 1 only: Anticancer hormonal treatment (except luteinizing hormone-releasing hormone [LHRH]) within 2 weeks before start of study intervention
* Part 1 only: Systemic anticancer therapy (except antibody-based anticancer therapy) or investigational agents within 3 weeks or 5 half-lives, whichever is longer
* Part 1 only: Antibody-based cancer therapy within 3 weeks before start of study intervention
* Part 1 only: Chloroquine/hydroxychloroquine within 2 weeks before start of study intervention
* Part 1 only: Clinically significant corneal disease
* Part 1 only: Has other uncontrolled or significant protocol-specified cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2030-02-14 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 44 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who experience an AE in the study will be presented.
Number of Participants Who Experience One or More Dose-Limiting Toxicities (DLTs) | Up to approximately 3 weeks
  A DLT is defined as any drug-related adverse event (AE) observed during the DLT evaluation period that meet pre-defined DTL criteria. Toxicities will be graded using National Cancer Institute Common Terminology for Adverse Events (NCI CTCAE) version 5.0, or the American Society for Transplant and Cellular Therapy (ASTCT) criteria. The number of participants who experience at least one DLT will be presented.
Number of Participants Who Discontinue Study Intervention Due to an AE | Up to approximately 44 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinue the study intervention due to an AE in the study will be presented.
Part 1: Objective Response Rate (ORR) | Up to approximately 44 months
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1). The percentage of participants who experience CR or PR as assessed by the investigator will be presented.

SECONDARY OUTCOMES:
Part 1, Part 2 (Arm 5 and Arm 6), and Part 3 (Arm 7): Duration of Response (DOR) | Up to approximately 44 months
  For participants who demonstrate a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by the investigator will be presented.
Part 1, Part 2 (Arm 6), and Part 3 (Arm 7): Progression-Free Survival (PFS) | Up to approximately 44 months
  PFS is defined as the time from randomization to the first documented PD or death due to any cause, whichever occurs first as assessed by RECIST 1.1. PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by the investigator will be presented.
Part 2 (Arm 5 and Arm 6) and Part 3 (Arm 7): ORR | Up to approximately 44 months
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1). The percentage of participants who experience CR or PR as assessed by the investigator will be presented.
Maximum Concentration (Cmax) of gocatamig | At designated timepoints (up to approximately 44 months)
  Cmax is the maximum concentration of the study drug observed in plasma. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine Cmax of the drug gocatamig.
Cmax of ifinatamab deruxtecan (I-DXd) | At designated timepoints (up to approximately 44 months)
  Cmax is the maximum concentration of the study drug observed in plasma. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine Cmax of the drug I-DXd.
Cmax of Anti-B7-H3 Antibody | At designated timepoints (up to approximately 44 months)
  Cmax is the maximum concentration of the study drug observed in plasma. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine Cmax of the anti-B7-H3 antibody.
Cmax of Deruxtecan (DXd) | At designated timepoints (up to approximately 44 months)
  Cmax is the maximum concentration of the study drug observed in plasma. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine Cmax of the drug payload deruxtecan (DXd).
Cmax of Durvalumab | At designated timepoints (up to approximately 44 months)
  Cmax is the maximum concentration of the study drug observed in plasma. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine Cmax of durvalumab.
Time to maximum concentration (Tmax) of gocatamig | At designated timepoints (up to approximately 44 months)
  Tmax is the amount of time that a drug is present at the maximum concentration is observed in plasma. Blood samples will be collected to determine the Tmax of the drug gocatamig.
Tmax of I-DXd | At designated timepoints (up to approximately 44 months)
  Tmax is the amount of time that a drug is present at the maximum concentration is observed in plasma. Blood samples will be collected to determine the Tmax of the drug I-DXd.
Tmax of Anti-B7-H3 Antibody | At designated timepoints (up to approximately 44 months)
  Tmax is the amount of time that the drug is present at the maximum concentration is observed in plasma. Blood samples will be collected to determine the Tmax of the anti-B7-H3 antibody.
Tmax of DXd | At designated timepoints (up to approximately 44 months)
  Tmax is the amount of time that the drug is present at the maximum concentration is observed in plasma. Blood samples will be collected to determine the Tmax of the drug payload DXd.
Area Under the Concentration-Time Curve Over the Dosing Interval t (AUCt) of gocatamig | At designated timepoints (up to approximately 44 months)
  AUCt is a measure of plasma drug concentration and time and is estimated as the area under the plot of plasma concentration against time after drug administration. Blood samples will be collected to determine the AUCt of the drug gocatamig.
AUCt of I-DXd | At designated timepoints (up to approximately 44 months)
  AUCt is a measure of plasma drug concentration and time and is estimated as the area under the plot of plasma concentration against time after drug administration. Blood samples will be collected to determine the AUCt of the drug I-DXd.
AUCt of Anti-B7-H3 Antibody | At designated timepoints (up to approximately 44 months)
  AUCt is a measure of plasma drug concentration and time and is estimated as the area under the plot of plasma concentration against time after drug administration. Blood samples will be collected to determine the AUCt of the anti-B7-H3 antibody.
AUCt of DXd | At designated timepoints (up to approximately 44 months)
  AUCt is a measure of plasma drug concentration and time and is estimated as the area under the plot of plasma concentration against time after drug administration. Blood samples will be collected to determine the AUCt of the drug payload Dxd.
Terminal Half-Life (t1/2) of gocatamig | At designated timepoints (up to approximately 44 months)
  t½ is defined as the time required for plasma drug concentration of study drug to decrease by 50% from peak. Blood samples will be collected to determine the t1/2 of the drug gocatamig.
t1/2 of I-DXd | At designated timepoints (up to approximately 44 months)
  t½ is defined as the time required for plasma drug concentration of study drug to decrease by 50% from peak. Blood samples will be collected to determine the t1/2 of the drug I-DXd.
t1/2 of Anti-B7-H3 Antibody | At designated timepoints (up to approximately 44 months)
  t½ is defined as the time required for plasma drug concentration of study drug to decrease by 50% from peak. Blood samples will be collected to determine the t1/2 of the anti-B7-H3 antibody.
t1/2 of DXd | At designated timepoints (up to approximately 44 months)
  t½ is defined as the time required for plasma drug concentration of study drug to decrease by 50% from peak. Blood samples will be collected to determine the t1/2 of the drug payload DXd.
Steady State Maximum Concentration (Cmax,ss) of gocatamig | At designated timepoints (up to approximately 44 months)
  Cmax,ss is a measure of the maximum level of drug in the blood, measured at steady state (time at which the amount of drug eliminated by the body is in equilibrium with the amount taken in). Blood samples will be collected to determine the Cmax,ss of the drug gocatamig.
Cmax,ss of I-DXd | At designated timepoints (up to approximately 44 months)
  Cmax,ss is a measure of the maximum level of drug in the blood, measured at steady state (time at which the amount of drug eliminated by the body is in equilibrium with the amount taken in). Blood samples will be collected to determine the Cmax,ss of the drug I-DXd.
Cmax,ss of Anti-B7-H3 Antibody | At designated timepoints (up to approximately 44 months)
  Cmax,ss is a measure of the maximum level of drug in the blood, measured at steady state (time at which the amount of drug eliminated by the body is in equilibrium with the amount taken in). Blood samples will be collected to determine the Cmax,ss of the anti-B7-H3 antibody.
Cmax,ss of DXd | At designated timepoints (up to approximately 44 months)
  Cmax,ss is a measure of the maximum level of drug in the blood, measured at steady state (time at which the amount of drug eliminated by the body is in equilibrium with the amount taken in). Blood samples will be collected to determine the Cmax,ss of the drug payload DXd.
Cmax,ss of Durvalumab | At designated timepoints (up to approximately 44 months)
  Cmax,ss is a measure of the maximum level of drug in the blood, measured at steady state (time at which the amount of drug eliminated by the body is in equilibrium with the amount taken in). Blood samples will be collected to determine the Cmax,ss of the durvalumab.
Steady State Ctrough (Ctrough,ss) of gocatamig | At designated timepoints (up to approximately 44 months)
  Ctrough,ss is defined as the trough concentration measured at steady state (time at which the amount of drug eliminated by the body is in equilibrium with the amount taken in). Blood samples will be collected to determine the Ctrough,ss of the drug gocatamig.
Ctrough,ss of I-DXd | At designated timepoints (up to approximately 44 months)
  Ctrough,ss is defined as the trough concentration measured at steady state (time at which the amount of drug eliminated by the body is in equilibrium with the amount taken in). Blood samples will be collected to determine the Ctrough,ss of the drug I-DXd.
Ctrough,ss of Anti-B7-H3 Antibody | At designated timepoints (up to approximately 44 months)
  Ctrough,ss is defined as the trough concentration measured at steady state (time at which the amount of drug eliminated by the body is in equilibrium with the amount taken in). Blood samples will be collected to determine the Ctrough,ss of the anti-B7-H3 antibody.
Ctrough,ss of DXd | At designated timepoints (up to approximately 44 months)
  Ctrough,ss is defined as the trough concentration measured at steady state (time at which the amount of drug eliminated by the body is in equilibrium with the amount taken in). Blood samples will be collected to determine the Ctrough,ss of the drug payload DXd.
Ctrough,ss of Durvalumab | At designated timepoints (up to approximately 44 months)
  Ctrough,ss is defined as the trough concentration measured at steady state (time at which the amount of drug eliminated by the body is in equilibrium with the amount taken in). Blood samples will be collected to determine the Ctrough,ss of durvalumab.
Steady State Time to Maximum Concentration (Tmax,ss) of gocatamig | At designated timepoints (up to approximately 44 months)
  Tmax,ss is the amount of time that a drug is present at the maximum concentration is observed in plasma measured at steady state (time at which the amount of drug eliminated by the body is in equilibrium with the amount taken in). Blood samples will be collected to determine the Tmax,ss of the drug gocatamig.
Tmax,ss of I-DXd | At designated timepoints (up to approximately 44 months)
  Tmax,ss is the amount of time that a drug is present at the maximum concentration is observed in plasma measured at steady state (time at which the amount of drug eliminated by the body is in equilibrium with the amount taken in). Blood samples will be collected to determine the Tmax,ss of the drug I-DXd.
Tmax,ss of Anti-B7-H3 Antibody | At designated timepoints (up to approximately 44 months)
  Tmax,ss is the amount of time that a drug is present at the maximum concentration is observed in plasma measured at steady state (time at which the amount of drug eliminated by the body is in equilibrium with the amount taken in). Blood samples will be collected to determine the Tmax,ss of the anti-B7-H3 antibody.
Tmax,ss of DXd | At designated timepoints (up to approximately 44 months)
  Tmax,ss is the amount of time that a drug is present at the maximum concentration is observed in plasma measured at steady state (time at which the amount of drug eliminated by the body is in equilibrium with the amount taken in). Blood samples will be collected to determine the Tmax,ss of the drug payload DXd.
Area Under the Steady State Concentration-Time Curve Over Dosing Interval t (AUCt,ss) of gocatamig | At designated timepoints (up to approximately 44 months)
  AUCt,ss is a measure of plasma drug concentration and time and is estimated as the area under the plot of plasma concentration against time after drug administration measured at steady state (time at which the amount of drug eliminated by the body is in equilibrium with the amount taken in). Blood samples will be collected to determine the AUCt,ss of the drug gocatamig.
AUCt,ss of I-DXd | At designated timepoints (up to approximately 44 months)
  AUCt,ss is a measure of plasma drug concentration and time and is estimated as the area under the plot of plasma concentration against time after drug administration measured at steady state (time at which the amount of drug eliminated by the body is in equilibrium with the amount taken in). Blood samples will be collected to determine the AUCt,ss of the drug I-DXd.
AUCt,ss of Anti-B7-H3 Antibody | At designated timepoints (up to approximately 44 months)
  AUCt,ss is a measure of plasma drug concentration and time and is estimated as the area under the plot of plasma concentration against time after drug administration measured at steady state (time at which the amount of drug eliminated by the body is in equilibrium with the amount taken in). Blood samples will be collected to determine the AUCt,ss of the anti-B7-H3 antibody.
AUCt,ss of DXd | At designated timepoints (up to approximately 44 months)
  AUCt,ss is a measure of plasma drug concentration and time and is estimated as the area under the plot of plasma concentration against time after drug administration measured at steady state (time at which the amount of drug eliminated by the body is in equilibrium with the amount taken in). Blood samples will be collected to determine the AUCt,ss of the drug payload DXd.
Steady state t1/2 (t1/2,ss) of gocatamig | At designated timepoints (up to approximately 44 months)
  t1/2,ss is defined as the time required for plasma drug concentration of study drug to decrease by 50% from peak measured at steady state (time at which the amount of drug eliminated by the body is in equilibrium with the amount taken in). Blood samples will be collected to determine the t1/2,ss of the drug gocatamig.
t1/2,ss of I-DXd | At designated timepoints (up to approximately 44 months)
  t1/2,ss is defined as the time required for plasma drug concentration of study drug to decrease by 50% from peak measured at steady state (time at which the amount of drug eliminated by the body is in equilibrium with the amount taken in). Blood samples will be collected to determine the t1/2,ss of the drug I-DXd.
t1/2,ss of Anti-B7-H3 Antibody | At designated timepoints (up to approximately 44 months)
  t1/2,ss is defined as the time required for plasma drug concentration of study drug to decrease by 50% from peak measured at steady state (time at which the amount of drug eliminated by the body is in equilibrium with the amount taken in). Blood samples will be collected to determine the t1/2,ss of the anti-B7-H3 antibody.
t1/2,ss of DXd | At designated timepoints (up to approximately 44 months)
  t1/2,ss is defined as the time required for plasma drug concentration of study drug to decrease by 50% from peak measured at steady state (time at which the amount of drug eliminated by the body is in equilibrium with the amount taken in). Blood samples will be collected to determine the t1/2,ss of the drug payload DXd.
Accumulation Ratio (AC) of gocatamig | At designated timepoints (up to approximately 44 months)
  Blood samples will be collected to determine the AC of the drug gocatamig.
AC of I-DXd | At designated timepoints (up to approximately 44 months)
  Blood samples will be collected to determine the AC of the drug I-DXd.
AC of Anti-B7-H3 Antibody | At designated timepoints (up to approximately 44 months)
  Blood samples will be collected to determine the AC of the anti-B7-H3 antibody.
AC of DXd | At designated timepoints (up to approximately 44 months)
  Blood samples will be collected to determine the AC of the drug payload DXd.
Incidence of Anti-Drug Antibodies (ADAs) Against gocatamig | At designated timepoints (up to approximately 44 months)
  Blood samples collected at designated timepoints will be used to determine the ADA response to gocatamig. The incidence of ADAs for gocatamig will be presented.
Incidence of ADAs Against I-DXd | At designated timepoints (up to approximately 44 months)
  Blood samples collected at designated timepoints will be used to determine the ADA response to I-DXd. The incidence of ADAs for I-DXd will be presented.
Incidence of ADAs Against Durvalumab | At designated timepoints (up to approximately 44 months)
  Blood samples collected at designated timepoints will be used to determine the ADA response to durvalumab. The incidence of ADAs for durvalumab will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (39):
- United States (9):
  - University of Colorado Anschutz Medical Campus ( Site 1110), Aurora, Colorado
  - University of Miami Hospital and Clinics, Sylvester Cancer Center ( Site 1111), Miami, Florida
  - University of Chicago ( Site 1108), Chicago, Illinois
  - Dana Farber Cancer Institute ( Site 1105), Boston, Massachusetts
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 1103), Hackensack, New Jersey
  - Roswell Park Cancer Institute ( Site 1107), Buffalo, New York
  - Providence Portland Medical Center ( Site 1101), Portland, Oregon
  - Sarah Cannon Research Institute ( Site 7001), Nashville, Tennessee
  - MEDICAL COLLEGE OF WISCONSIN ( Site 1112), Milwaukee, Wisconsin
- Princess Alexandra Hospital ( Site 5300), Wooloongabba, Queensland, Australia
- Chile (2):
  - FALP ( Site 2100), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 2101), Santiago, Region M. de Santiago
- China (6):
  - Beijing Cancer Hospital ( Site 5401), Beijing, Beijing Municipality
  - Fujian Cancer Hospital ( Site 5413), Fuzhou, Fujian
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School-Oncology ( Site 5403), Nanjing, Jiangsu
  - Shanghai Chest Hospital ( Site 5400), Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital ( Site 5405), Shanghai, Shanghai Municipality
  - The First Affiliated Hospital, Zhejiang University ( Site 5404), Hangzhou, Zhejiang
- Israel (4):
  - Rambam Health Care Campus ( Site 3202), Haifa
  - Shaare Zedek Medical Center ( Site 3200), Jerusalem
  - Rabin Medical Center ( Site 3203), Petah Tikva
  - Sheba Medical Center ( Site 3201), Ramat Gan
- Japan (4):
  - Aichi Cancer Center ( Site 5000), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 5001), Kashiwa, Chiba
  - Kansai Medical University Hospital ( Site 5004), Hirakata, Osaka
  - Cancer Institute Hospital of JFCR ( Site 5002), Koto, Tokyo
- South Korea (2):
  - Seoul National University Hospital ( Site 5100), Seoul
  - Samsung Medical Center ( Site 5101), Seoul
- Spain (7):
  - HOSPITAL CLÍNIC DE BARCELONA ( Site 3310), Eixample, Barcelona
  - Institut Català d'Oncologia - L'Hospitalet ( Site 3317), L'Hospitalet de Llobregat, Barcelona
  - Hospital Clinico San Carlos... ( Site 3316), Madrid, Madrid, Comunidad de
  - Hospital Universitari Vall d'Hebron ( Site 3311), Barcelona
  - Hospital Universitario Fundación Jiménez Díaz-START Madrid-FJD ( Site 3315), Madrid
  - Hospital Universitario HM Sanchinarro ( Site 3313), Madrid
  - Hospital Universitario Virgen de la Victoria ( Site 3312), Málaga
- Taiwan (2):
  - National Cheng Kung University Hospital ( Site 5202), Tainan
  - Taipei Medical University Hospital ( Site 5201), Taipei
- Turkey (Türkiye) (2):
  - Hacettepe Universite Hastaneleri ( Site 3410), Ankara
  - Ankara Bilkent Sehir Hastanesi ( Site 3412), Ankara

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com